CLINICAL TRIAL: NCT07128784
Title: The Impact of Aerobic Exercise Training on Cardiopulmonary Exercise Capacity in Patients With Heart Failure
Brief Title: Aerobic Training and Cardiopulmonary Responses In Heart Failure
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: TABED 2-25-1203
Record Dates: First submitted 2025-06-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Cardiopulmonary Exercise Test; Aerobic Capacity; Aerobic Exercise
Keywords: cardiopulmonary exercise test; aerobic capacity; aerobic exercise; heart failure
MeSH Terms: conditions — Heart Failure | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- aerobic exercise
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — continuous, moderate intencity aerobic exercise, 3 days a week, 30 minutes per day, 150/min per week for a total of 6 weeks

SUMMARY:
The goal of this observational study is to learn about the short-term effects of aerobic exercise in heart failure patients who were given exercise prescription with cardiopulmonary exercise stres test acocording to aerobic capacity . The main question it aims to answer is:

Does aerobic exercise increase aerobic capacity and quality of life Participants already taking aerobic capacity as part of their regular medical care for Heart failure will asses with cardiopulmonary exercise test and clinical questionaries about quality of life and depression-anxiety level before and after aerobic exercise treatment .

DETAILED DESCRIPTION:
The goal of this observational study is to learn about the short-term effects of aerobic exercise in heart failure patients who were given exercise prescription with cardiopulmonary exercise stres test acocording to aerobic capacity . The main question it aims to answer is:

Does aerobic exercise increase aerobic capacity and quality of life Participants already taking aerobic capacity as part of their regular medical care for Heart failure will asses with cardiopulmonary exercise test and clinical questionaries about quality of life and depression-anxiety level before and after aerobic exercise treatment .

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75,
* Diagnosed with compensated HF,
* BMI 18-30 kg/m²,
* LVEF < 0.4,
* NYHA 2-3,
* Clinical symptoms have been stable for at least 2 weeks, and the dose of angiotensin-converting enzyme inhibitor/angiotensin receptor antagonist/angiotensin receptor inhibitor, beta-blocker, aldosterone inhibitor, and other drugs has been stable for at least 2 weeks.

Exclusion Criteria:

* History of a heart implant device within the last 6 weeks or a heart implant device or heart transplant plan within the next 12 months,
* Acute coronary syndrome within the last 6 weeks, severe valvular heart disease, congenital heart disease, severe hypertrophic obstructive cardiomyopathy, acute myocarditis/pericarditis, intracardiac thrombosis, primary pulmonary hypertension,
* Uncontrolled hypertension (systolic blood pressure >200 mmHg and/or diastolic blood pressure >110 mmHg),
* Severe arrhythmias such as ventricular tachycardia, frequent multisource premature ventricular beats, high atrioventricular block, and significant QT interval prolongation during exercise testing,
* Progressive dyspnea or
* Loss of exercise endurance at rest within the last 3-5 days under low-intensity exercise load (<2 MET) who have suffered myocardial ischemia,
* Patients with cognitive impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-75 age of years , male and female , diagnosed with heart failure with reduced EF
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
cardiopulmonary exercise test results | 6 weeks
  Cardiovascular responses: VO2 max value (ml/kg/dk)
cardiopulmonary exercise test results | 6 weeks
  Cardiovascular responses: heart rate (bpm, beats/min)
cardiopulmonary exercise test results | 6 weeks
  gas exchange response: VE/VCO2: EQCO2: Ventilatory equivalent for carbon dioxide minute ventilation while the produced CO₂ is removed,
cardiovascular exercise test result: Gas exchange parameters: | 6 weeks
  PETCO₂ (partial end-tidal carbon dioxide), kilopascal

SECONDARY OUTCOMES:
Short Form (36) Health Scale | 6 weeks
  Short Form (36) Health Scale
  Description:
  The SF-36 is a widely used, patient-reported survey of health status designed to assess overall health-related quality of life. It evaluates physical and mental health across multiple dimensions and is commonly used in clinical research and health outcomes studies.
  Domains Assessed (8 Subscales): Physical Functioning , Role Limitations due to Physical Health,Pain, General Health Perceptions Vitality, Social Functioning, Role Limitations due to Emotional Problems, Mental Health
  These can also be summarized into two main component scores:
  Physical Component Summary (PCS) Mental Component Summary (MCS)
  Scoring Range:
  Each subscale is scored from 0 to 100. 0 represents the worst possible health status; 100 represents the best possible health status.
  Interpretation of Scores:
  Higher scores indicate better health outcomes and higher quality of life, lower scores reflect poorer perceived healt
Hospital Anxiety and Depression Scale | 6 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment tool developed to detect states of anxiety and depression in patients in non-psychiatric hospital clinics. It is widely used in both clinical practice and research settings to screen for emotional distress, especially in individuals with physical illnesses.
  Structure:
  The scale consists of 14 items, divided into two subscales:
  HADS-A (Anxiety) - 7 items HADS-D (Depression) - 7 items Each item assesses symptoms experienced over the past week.
  Scoring Range:
  Each item is scored from 0 to 3. Subscale scores range from 0 to 21 for both anxiety and depression.
  Interpretation of Scores (per subscale):
  0-7: Normal 8-10: Borderline abnormal (mild) 11-21: Abnormal (clinically significant)
  Direction of Scores:
  Higher scores indicate greater severity of anxiety or depression symptoms. Lower scores suggest fewer or no symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lelonek M. Heart failure with preserved ejection fraction after the PARAGON-HF trial results: current knowledge and future directions. Kardiol Pol. 2020 Dec 23;78(12):1199-1205. doi: 10.33963/KP.15639. Epub 2020 Oct 6. PMID 33021355
- [Background] Conrad N, Judge A, Tran J, Mohseni H, Hedgecott D, Crespillo AP, Allison M, Hemingway H, Cleland JG, McMurray JJV, Rahimi K. Temporal trends and patterns in heart failure incidence: a population-based study of 4 million individuals. Lancet. 2018 Feb 10;391(10120):572-580. doi: 10.1016/S0140-6736(17)32520-5. Epub 2017 Nov 21. PMID 29174292